CLINICAL TRIAL: NCT04547894
Title: A Study to Evaluate the Pharmacokinetics of ASC09F in Healthy Subjects After Multiple Doses
Brief Title: A Study of the Pharmacokinetics of ASC09F in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Beijing YouAn Hospital (Other)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-ASC09F-I-CTP-01
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASC09F (Experimental): ASC09F one tablet at a time, once per day, up to 7 days.
  Interventions: Drug: ASC09F

INTERVENTIONS:
Drug: ASC09F — ASC09F (300 mg ASC09 and 100 mg Ritonavir) one tablet at a time, once per day, up to 7 days.

SUMMARY:
The objective of this study is to evaluate the pharmacokinetic parameters of ASC09F in healthy subjects after multiple oral dosing.

DETAILED DESCRIPTION:
This study will evaluate the safety and the pharmacokinetics of ASC09F tablets in healthy volunteers. Subjects will receive 7 days multiple oral doses of ASC09F tablets.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-45 (including boundary value), half men and half women. 2. Male weight ≥ 50kg, female weight ≥ 45kg;BMI ranges from 19 to 30kg/m2 (boundary value included).

  3. According to the medical history, physical examination, vital signs, laboratory examination and 12 lead electrocardiogram (ECG) examination, the general health condition is good, and there is no clinically significant abnormality in each index.

  4. Unplanned pregnancy within half a year and willing to take effective contraceptive measures within 30 days from the first administration of the study drug to the last administration.

  5. The pregnancy test of female subjects during the screening period is negative.

  6. Those who voluntarily sign the informed consent.

Exclusion Criteria:

* 1. Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCV Ab), HIV antibody (HIV Ab) and syphilis antibody were tested positive.

  2. People who have taken special diet (including carambola, dragon fruit, mango, grapefruit, orange, etc.) or drunk alcohol, or had strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion within 2 weeks before taking the study drug.

  3. Heavy smokers (14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 mL wine;Smoking daily ≥ 5 sticks) and no smoking or alcohol prohibition during the study period.

  4. Ingesting chocolate, any food or drink containing caffeine or xanthine in the 24 hours prior to taking the study drug.

  5. Patients who had donated blood or lost blood of more than 400ml within 3 months before taking the study drug.

  6. Those who have participated in other clinical trials and received study drug treatment within 3 months before taking study drug.

  7. Alcoholic or nonalcoholic fatty liver disease. 8. In addition to the above, the researchers judge that the participants are not suitable to participate in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
AUC of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Area under the plasma concentration versus time curve after
Cmax of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Peak Plasma Concentration after single and multiple oral doses of ASC09F administered to Chinese healthy volunteers.

SECONDARY OUTCOMES:
t1/2 of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Terminal-Phase Half-Life after single and multiple oral doses of ASC09F administered to Chinese healthy volunteers volunteers.
CL/F of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Apparent Systemic Clearance after single and multiple oral dose of ASC09F administered to Chinese healthy volunteers.
Vd/F of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Apparent Volume of Distribution after single and multiple oral dose of ASC09F administered to Chinese healthy volunteers.
Evaluation of the safety of ASC09F in healthy volunteers | Up to 11 days
  Evaluate number of adverse events as a measure of safety of ASC09F.
Tmax of ASC09F | On Day 1,2,3,4 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 11 days.
  Evaluate the Time to reach the maximum plasma concentration after single single and multiple oral doses of ASC09F administered to Chinese healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dierynck I, Van Marck H, Van Ginderen M, Jonckers TH, Nalam MN, Schiffer CA, Raoof A, Kraus G, Picchio G. TMC310911, a novel human immunodeficiency virus type 1 protease inhibitor, shows in vitro an improved resistance profile and higher genetic barrier to resistance compared with current protease inhibitors. Antimicrob Agents Chemother. 2011 Dec;55(12):5723-31. doi: 10.1128/AAC.00748-11. Epub 2011 Sep 6. PMID 21896904
- [Background] Hoetelmans RM, Dierynck I, Smyej I, Meyvisch P, Jacquemyn B, Marien K, Simmen K, Verloes R. Safety and pharmacokinetics of the HIV-1 protease inhibitor TMC310911 coadministered with ritonavir in healthy participants: results from 2 phase 1 studies. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):299-305. doi: 10.1097/QAI.0000000000000011. PMID 24121757
- [Background] Stellbrink HJ, Arasteh K, Schurmann D, Stephan C, Dierynck I, Smyej I, Hoetelmans RM, Truyers C, Meyvisch P, Jacquemyn B, Marien K, Simmen K, Verloes R. Antiviral activity, pharmacokinetics, and safety of the HIV-1 protease inhibitor TMC310911, coadministered with ritonavir, in treatment-naive HIV-1-infected patients. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):283-9. doi: 10.1097/QAI.0000000000000003. PMID 24121756